CLINICAL TRIAL: NCT03809611
Title: A 3-month, Randomized, Placebo-controlled, Double-masked, Multi-center Study to Evaluate the Safety and Efficacy of Topical Ocular UNR844-Cl in Subjects With Presbyopia
Brief Title: A Study of Safety and Efficacy of UNR844 Chloride (UNR844-Cl) Eye Drops in Subjects With Presbyopia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUNR844A2203
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Results first posted 2020-11-27 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Presbyopia
Keywords: Presbyopia, adults, randomized study, placebo
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-mask(Investigator, patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UNR844-Cl Ophthalmic Solution (Experimental): 1.5% UNR844-Cl ophthalmic solution for twice-daily dosing
  Interventions: Drug: UNR844-Cl
- Placebo Ophthalmic Solution (Placebo Comparator): placebo ophthalmic solution for twice-daily dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UNR844-Cl — 1.5% Ophthalmic solution for topical ocular administration
  Other Names: Lipoic acid choline ester chloride, EV06
  Arms: UNR844-Cl Ophthalmic Solution
Drug: Placebo — placebo
  Other Names: Vehicle
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The purpose of this study was to assess the effect of topical UNR844-Cl (lipoic acid choline ester chloride) ophthalmic solution on near visual function in presbyopic subjects.

DETAILED DESCRIPTION:
This was a multi-center, double-masked, placebo-controlled, randomized, parallel-group study. The total duration of the study was approximately 3 months. Approximately 120 presbyopic subjects were to be enrolled into the study.

Presbyopic subjects aged 45 to 55 years were the primary age group in this study.

Screening and Baseline: Subjects were screened for eligibility followed by a baseline visit after which they were randomized to receive either UNR844-Cl (1.5%, equivalent to 1.3% freebase) or Placebo, dosed one drop in each eye twice daily, for 3 months.

Randomized subjects attended the following study visits after baseline: at Week 2, Month 1, Month 2 and Month 3.

The primary objective of this study was to assess the efficacy of UNR844-Cl on binocular distance corrected near visual acuity (DCNVA) in presbyopic subjects aged 45 to 55 years with the primary endpoint being the change from baseline in binocular DCNVA in subjects aged 45 to 55 years at Month 3 after UNR844-Cl or Placebo treatment.

There were two secondary endpoints:

1. To assess the efficacy of UNR844-Cl on achieving 75 or more Early Treatment Diabetic Retinopathy Study (ETDRS) letters in binocular DCNVA in presbyopic subjects aged 45 to 55 years with endpoint being the proportion of subjects aged 45 to 55 years achieving 75 or more ETDRS letters in binocular DCNVA at Month 3 after UNR844-Cl or Placebo treatment.
2. To assess the safety of UNR844-Cl in presbyopic subjects by the frequency of treatment emergent adverse events (AEs) and treatment emergent serious adverse events (SAEs) in all subjects after UNR844-Cl or Placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Impaired near vision in each eye and when using both eyes, without any near correction
* Need a certain level of near correction

Exclusion Criteria:

* Impaired distance vision in either eye, with distance correction (if any)
* Severe short- or long-sightedness
* Any significant medical or clinical conditions affecting vision, the eyes or general health

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (13):
  - Novartis Investigative Site, Mission Hills, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Mt. Dora, Florida
  - Novartis Investigative Site, Washington, Missouri
  - Novartis Investigative Site, Allenwood, Pennsylvania
  - Novartis Investigative Site, Cranberry Township, Pennsylvania
  - Novartis Investigative Site, Kingston, Pennsylvania
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Cedar Park, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
URL: https://www.clinicalstudydatarequest.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- UNR844-Cl: 1.5% UNR844-Cl
- Placebo Ophthalmic Solution: placebo
Period: Overall Study
Arm/Group | UNR844-Cl | Placebo Ophthalmic Solution
Started | 62 | 62
Completed | 61 | 61
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UNR844-Cl | Placebo Ophthalmic Solution | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (4.97) | 54.2 (5.01) | 54.1 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 22 | 21 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 8 | 15
  White | 50 | 51 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Binocular Distance-corrected Near Visual Acuity (DCNVA) From Baseline
Description: Change from baseline in binocular DCNVA in subjects aged 45 to 55 years at Month 3 after UNR844-Cl or placebo treatment. Low contrast (10% contrast) DCNVA at 40 cm is measured binocularly using an electronic visual acuity testing system. This assessment was performed with subjects corrected for any distance refractive errors. The system provided distance-corrected low contrast near visual acuity in an Early Treatment Diabetic Retinopathy Study (ETDRS) letter numerical score. High monocular DCNVA ETDRS letter scores represent good vision; Low monocular DCNVA ETDRS letter scores represent poor vision.
Time Frame: Baseline and at Month 3
Population: All randomized subjects aged 45 to 55 years at baseline
Measure: Least Squares Mean (Standard Error); unit: number of letters read correctly
Arm/Group | UNR844-Cl | Placebo Ophthalmic Solution
Number analyzed (Participants) | 40 | 38
number of letters read correctly | 6.1 (1.24) | 4.5 (1.27)
Statistical Analysis 1: Comparison: UNR844-Cl vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.1832, Mixed Models Analysis — One-sided p-value for treatment difference; Mean Difference (Net) = 1.6, 90% CI 2-sided [-1.34 to 4.56], Standard Error of Mean 1.77

2. Secondary Outcome: Number and Percentage of Subjects Aged 45 to 55 Years Achieving 75 or More Early Treatment Diabetic Retinopathy Study (ETDRS) Letters in Binocular DCNVA at Month 3
Description: as for outcome 1
Time Frame: month 3
Population: l randomized subjects aged 45 to 55 years at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | UNR844-Cl | Placebo Ophthalmic Solution
Number analyzed (Participants) | 40 | 38
Participants | 10 | 6
Statistical Analysis 1: Comparison: UNR844-Cl vs Placebo Ophthalmic Solution; Test type: Superiority; p = 0.2830, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.9, 90% CI 2-sided [0.72 to 4.78]

3. Secondary Outcome: Number of Subjects With Adverse Events, Ocular Adverse Events, Deaths, Other Serious Adverse Events, or Adverse Events Leading to Study Drug Discontinuation
Description: Frequency of treatment emergent adverse events and treatment emergent serious adverse events in all subjects. Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 120 days.
Time Frame: 4 months
Population: All randomized and treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | UNR844-Cl | Placebo Ophthalmic Solution
Number analyzed (Participants) | 62 | 62
Participants
  Any adverse events (AEs) | 14 | 5
  Any ocular adverse events | 4 | 4
  Any non-ocular adverse events | 11 | 2
  Any severe adverse events | 0 | 0
  Any ocular severe adverse events | 0 | 0
  Any non-ocular severe adverse events | 0 | 0
  Any study drug related adverse events | 4 | 1
  Any study drug related ocular adverse events | 0 | 1
  Any study drug related non-ocular adverse events | 4 | 0
  Any adverse events leading to study drug disc. | 0 | 0
  Any ocular AEs leading to study drug disc. | 0 | 0
  Any non-ocular AEs leading to study drug disc. | 0 | 0
  Any serious adverse events | 0 | 0
  Any ocular serious adverse events | 0 | 0
  Any non-ocular serious adverse events | 0 | 0
  Any study drug related serious adverse events | 0 | 0
  Any study drug related ocular serious AEs | 0 | 0
  Any study drug related non-ocular serious AEs | 0 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 120 days.
Groups:
- UNR844-Cl: UNR844-Cl
- Total: Total
Arm/Group | UNR844-Cl | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62 | 0/124
Other Adverse Events (participants affected / at risk) | 14/62 | 5/62 | 19/124
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UNR844-Cl (N=62) | Placebo (N=62) | Total (N=124)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 1
Lenticular opacities (Eye disorders) | 0 | 1 | 1
Visual impairment (Eye disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Instillation site pain (General disorders) | 0 | 1 | 1
Sensation of foreign body (General disorders) | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vital dye staining cornea present (Investigations) | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 0 | 3
Headache (Nervous system disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03809611/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03809611/SAP_001.pdf